CLINICAL TRIAL: NCT07278050
Title: Interscalene Block vs Serratus Posterior Superior Intercostal Plane Block on Postoperative Analgesia Management After Arthroscopic Shoulder Surgery: A Randomized Prospective Study
Brief Title: Interscalene Block vs Serratus Posterior Superior Intercostal Plane Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-1405
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Pain; Shoulder Disease
Keywords: Arthroscopic Shoulder Surgery; Postoperative analgesia management; serratus posterior superior intercostal plane block; Interscalene brachial plexus block
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is the serratus posterior superior intercostal plane block group. The second one is an interscalene brachial plexus block.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SPSIPB = SPSIPB group (Active Comparator): SPSIPB will be performed
  Interventions: Drug: Serratus posterior superior intercostal plane block; Drug: Postoperative analgesia management
- Group ESPB = ESPB group (Active Comparator): ESPB will be performed
  Interventions: Drug: Erector spinae plane block; Drug: Postoperative analgesia management

INTERVENTIONS:
Drug: Erector spinae plane block — The procedure will be performed with the patient in the supine position after surgery before extubation. ESPB will be performed. The US probe will be placed longitudinally 2-3 cm lateral to the T2 transverse process. The erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle will be inserted in a caudo-cranial direction, and then, for correction, 5 ml of saline will be injected deep into the erector spinae muscle fascia. Following confirmation of the correct position of the needle, 30 mL %0.25 bupivacaine will be administered for the block.
  Arms: Group ESPB = ESPB group
Drug: Serratus posterior superior intercostal plane block — A high-frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The procedure will be performed with the patient in the sitting position after surgery before extubation. After the scapula is shifted slightly laterally, the US probe is placed sagittal at the upper corner of the spina scapula, and the serratus posterior superior muscle is visualized with the third rib. The in-plane technique will be used. The block needle will be advanced in the craniocaudal direction to enter between the serratus posterior superior and the third rib. The block location will be confirmed by injecting 5 ml of saline between the rib and the muscle. After the block location is confirmed, 30 ml of 0.25% concentration bupivacaine will be used.
  Arms: Group SPSIPB = SPSIPB group
Drug: Postoperative analgesia management — Patients will be administered ibuprofen 400 mg IV every 8 hours in the postoperative period. A patient-controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol including a 10 mcg bolus without an infusion dose, a 10-minute lockout time, and a 4-hour limit. If the NRS score is ≥ 4, 0.5 mg kg-1 IV meperidine will be administered as a rescue analgesic. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.

SUMMARY:
Postoperative pain is important following arthroscopic shoulder surgery. Postoperative effective pain treatment provides early mobilization and a shorter hospital stay. Ultrasound (US)-guided brachial plexus blocks, such as interscalene and supraclavicular block, are usually performed. Interscalen brachial plexus block (ISCB) is one of the most preferred techniques among these.

Ultrasound (US) guided serratus posterior superior block (SPSPB) is a new interfacial plane block defined by Tulgar et al in 2023. It is based on injection on the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in conditions such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. The SPS muscle is located at the C7-T2 level. It attaches to the lateral edges of the second and fifth ribs. It is innervated by the lower cervical and upper intercostal nerves. With the SPS block, these nerves are blocked, and analgesia is provided. It has been reported that SPSIPB provides effective analgesia after shoulder surgery.

The aim of this study is to compare the efficacy of the US-guided SPSIPB and ISCB for postoperative analgesia management after arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
Postoperative pain is an important issue in patients who have undergone arthroscopic shoulder surgery. Pain causes a few problems: uncomfortable patients, negative outcomes, and longer rehabilitation. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization, such as infection and thromboembolism, may be reduced. Various techniques may be used for postoperative pain treatment. Opioids are one of the most preferred drugs among analgesic agents. Parenteral opioids are generally administered to patients after surgery. However, opioids have undesirable adverse events such as nausea, vomiting, itching, sedation, and respiratory depression (opioid-related adverse events).

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment following arthroscopic shoulder surgery. Ultrasound (US)-guided brachial plexus blocks, such as interscalene and supraclavicular block, are commonly used. Interscalen brachial plexus block (ISCB) is one of the most preferred techniques among these.

US-guided interfascial plane blocks have been used increasingly due to the advantages of ultrasound in anesthesia practice. Ultrasound (US) guided serratus posterior superior block (SPSPB) is a new interfacial plane block defined by Tulgar et al in 2023. It is based on injection on the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in conditions such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. The SPS muscle is located at the C7-T2 level. It attaches to the lateral edges of the second and fifth ribs. It is innervated by the lower cervical and upper intercostal nerves. With the SPS block, these nerves are blocked, and analgesia is provided.

In the cadaveric study of Tulgar et al., it was determined that the spread of the serratus posterior superior interfacial plane block, 7-10 intercostal levels on the left side, only in the superficial fascia of the trapezius muscle. Spread dye was observed at intercostal levels, absent on the right. There was prominent staining on both sides of the deep trapezius muscle. Both the surface and skin of the rhomboid major were stained, while the rhomboid minor was only stained in the skin. SPSP block will provide successful analgesia in procedures involving the thoracic region, such as chronic myofascial pain, breast surgery, thoracic surgery, and shoulder surgery. There is no randomized study in the literature evaluating the effectiveness of the SPSP block for postoperative analgesia management after shoulder surgery.

This study aims to compare the efficacy of the US-guided SPSIPB and ISCB for postoperative analgesia management after arthroscopic shoulder surgery. The primary aim is to compare postoperative opioid consumption (fentanyl), and the secondary aim is to evaluate postoperative pain scores (NRS), adverse effects related to opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for arthroscopic shoulder surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption (fentanyl) | Change from baseline opioid consumption at postoperative 1, 2, 4, 8, 16, 24 hours
  The primary aim is to compare postoperative opioid consumption

SECONDARY OUTCOMES:
Pain scores (Numerical rating scores-NRS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16 and 24 hours
  The secondary aim is to compare NRS at the postoperative 24 h. Postoperative pain assessment will be performed using the NRS (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded
Need for rescue analgesia (meperidine) | Postoperative 24 hours period
  The secondary aim is to compare rescue analgesia used in the postoperative 24 h.
Adverse events | Postoperative 24 hours period
  The secondary aim is to compare the adverse events (nausea, vomiting, itching) related to opioid use

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Ciftci B, Alver S, Ahiskalioglu A, Bilal B, Tulgar S. Serratus posterior superior intercostal plane block: novel thoracic paraspinal block for thoracoscopic and shoulder surgery. Minerva Anestesiol. 2024 Apr;90(4):345-347. doi: 10.23736/S0375-9393.23.17827-8. Epub 2024 Jan 19. No abstract available. PMID 38240640
- [Background] Kapukaya F, Ekinci M, Ciftci B, Atalay YO, Golboyu BE, Kuyucu E, Demiraran Y. Erector spinae plane block vs interscalene brachial plexus block for postoperative analgesia management in patients who underwent shoulder arthroscopy. BMC Anesthesiol. 2022 May 12;22(1):142. doi: 10.1186/s12871-022-01687-5. PMID 35550031
- [Background] Zhang Y, Li H, Xu S, Guo R, Ma D, Wang Y. Understanding the Anatomy of Posterior Cervical Interfascial Space: Implications for Regional Blocks and Pain Management. A Narrative Review. Pain Ther. 2025 Aug;14(4):1203-1222. doi: 10.1007/s40122-025-00754-2. Epub 2025 Jun 16. PMID 40522591
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093